CLINICAL TRIAL: NCT05132179
Title: A Randomized Double-blind Clinical Trial Comparing Hypochlorous Acid and Polyhexamethylene Biguanide in Treating Diabetic Foot Ulcers
Brief Title: Treating Diabetic Foot Ulcers, Comparing Two Topical Antimicrobial Agents, Dakin´s and Prontosan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Marcus Lind, Professor, consultant Endocrinology, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0011365-36
Record Dates: First submitted 2021-09-24; First posted 2021-11-24 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer, DFU; Healing; Dakin´s solution; Prontosan Wound Irrigation Solution; Antibiotic consumption; Healing pattern; Microbiological variables; Cost-effectiveness; Diabetes type 1 and 2; Topical antimicrobial agent; Hypochlorous Acid; PHMB; Topical treatment
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 1 | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled, multi-center, clinical trial with parallel-group design
Who Masked: Participant, Care Provider, Investigator
Masking Description: The wound irrigation solutions will be filled in identical 5 ml syringes, marked with study number and date of filling. To mask the smell of chlorine a tin without lid with 15 ml 5% chloride will be placed maximally 1 meter from the treating place
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOCl arm (Active Comparator): Dakin´s Solution, with the active substance Hypochlorous Acid, HOCl was first invented 1915 for use on infected war wounds. The DFU will be cleaned with HOCl twice a week. The treatment will be performed in accordance with instructions for Prontosan, PHMB.
  Interventions: Drug: Dakins Full Strength Solution, 0.5% Topical Solution, HOCl solution
- PHMB arm (No Intervention): Prontosan, with the active substance PHMB, is recommended by 19 out of 21 regions in Sweden, for cleaning DFU. The DFU will be cleaned with PHMB twice a week. The treatment will be performed in accordance with instructions for Prontosan, PHMB.

INTERVENTIONS:
Drug: Dakins Full Strength Solution, 0.5% Topical Solution, HOCl solution — Dakin´s solution is a 50/50 mixture of 1% sodiumhypochlorite and 2% sodiumhydrocarbonate, the mixture is a 0,5% chlorine solution. Dakin´s solution is not used in Sweden on wound. Dakin´s solution is only used in dental care in Sweden.
  Other Names: Dakins
  Arms: HOCl arm

SUMMARY:
202 Diabetic foot ulcers will be cleaned with either Hypochlorous Acid, HClO or Polyhexamethylene biguanide, PHMB twice a week until healed or 24 weeks. Primary objective is to find out if cleaning DFU with HClO is more effective in obtaining complete healing than PHMB.

DETAILED DESCRIPTION:
202 persons with diabetes and diabetic foot ulcers, DFU will be randomized to treatment with either Hypochlorous Acid, HClO or Polyhexamethylene biguanide, PHMB. The study is double blind and controlled. The cleaning will be done as instruction for PHMB, twice a week until complete healing of the DFU or if not healed 24 weeks. Complete healing is defined as intact skin covering the place where there was an ulcer. Primary objective is time to healing, if cleaning DFU with HClO is more effective in obtaining complete healing of DFU than PHMB. Secondary objectives are to examine if HClO compared with PHMB differ when treating DFU with respect to: a. Proportion of DFU that heals within 12 weeks of treatment, b. The size of the DFU´s surface area over 24 weeks of treatment, c. The depth of the DFU over 24 weeks d. The use of antibiotics over 24 weeks of treatment, e. The quality of life using EQ-5D questionnaire. Explorative objectives are to examine if HClO compared with PHMB differ when treating DFU with respect to: a. Change in healing pattern (sub study in Västra Götaland), b. Change in microbiological variables (sub study in Västra Götaland), c. The quality of life using SF-12 questionnaire, d. Cost effectiveness and other health-economical aspects

ELIGIBILITY:
Inclusion Criteria: Informed consent obtained before trial-related activities,

* Diabetes Mellitus type 1 or 2 or due to pancreatitis
* Foot ulcer since 3 weeks or more
* Ulcer surface area 9 mm2 or more
* Age 18 years old or more

Exclusion Criteria:

* Persons in need of intensive care or dialysis
* Persons in need of vascular intervention, critically impaired circulation (toe-pressure < 30 mm Hg)
* Event of myocardial infarction or stroke during the last three months
* Debut of atrial fibrillation or heart failure during the last three months
* Current treatment of malignancy
* Treatment with corticosteroids with a dose corresponding to 50 mg Prednisolon
* Severe wound infection according to International Working Group of Diabetic Foot, IWGDF at least two of following signs: body temperature <36 C or >38 C, heart rate >90/minute, respiration rate >20/minute, LPK >12x10^9/L
* Planned changed residence in the coming 12 months requiring change of clinic for wound treatment during the follow-up time
* Age under 18 years old
* Diabetes of MOODY type
* Current known pregnancy or planned pregnancy next 26 weeks
* Participation in another clinical trial evaluating any treatment
* Other reasons judged by the investigator that the patient is unsuitable for participation in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to healing | 24 weeks
  The primary efficacy analysis of difference in time to healing from randomisation up to 24 weeks between the two randomised groups. Analysis will be performed using Cox regression. The healing date will be defined as the first visit when the ulcer is fully covered with skin.

SECONDARY OUTCOMES:
Proportion of DFU that heals within 12 weeks of treatment | 12 weeks
  Difference in proportion healed DFU between groups at week 12 will be estimated using Fisher´s exact test
Change of DFU´s surface area | 24 weeks
  The size of surface area measured with a mm ruler in photo of the DFU. The surface area of The DFU will be measured weekly for 24 weeks or until healed from weekly photo with a mm ruler in the photo. The calculation of the area will be done by a person not involved in the treatment. For each participants and time point, the percentage change of the ulcer size (area and volume) will be calculated in relation to randomisation. For each group (HOCl and PHMB, respectively), the average change in ulcer size (area and volume) will be calculated, whereafter any difference between the two groups will be examined for statistical significance.
Change of diabetic foot ulcer´s, DFU´s, depth | 24 weeks
  The depth of diabetic foot ulcer measured with digital pair of calipers weekly for 24 weeks or until healed. For each participant and time point, the percentage change of the ulcer size (area and volume) will be calculated in relation to the date of randomisation. For each group (HOCl and PHMB, respectively), the average change in ulcer size (area and volume) will be calculated, whereafter any difference between the two groups will be examined for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, Prof, Principal Investigator — University of Gothenburg, Sahlgrenska Academy
Locations (1):
- NU sjukvarden, Uddevalla, Trollhattan, Sweden